CLINICAL TRIAL: NCT02722941
Title: Evaluation of Panobinostat (LBH589) as Maintenance Therapy in Multiple Myeloma Following Autologous Hematopoietic Cell Transplantation
Brief Title: Panobinostat (LBH589): Multiple Myeloma - Autologous Hematopoietic Cell Transplantation (HCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18430; CLBH589DUS97T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: autologous hematopoietic cell transplant (HCT); autologous
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Maintenance Therapy (Active Comparator): Panobinostat (LBH589): 20 mg by mouth three (3) times per week, every other week, of a 28-day schedule.
  Interventions: Drug: Panobinostat
- Cohort B: Maintenance Therapy (Active Comparator): Panobinostat (LBH589): 10 mg by mouth daily for seven (7) days, every other week, of a 28-day schedule.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Maintenance therapy dosing as outlined in Cohorts A and B.
  Other Names: LBH589

SUMMARY:
The purpose of this study is to learn more about ways to prevent or delay relapse of multiple myeloma (MM). This study will determine the best dosing schedule of LBH589 maintenance therapy as well as the safety (side effects) and tolerability of LBH589 maintenance therapy after autologous hematopoietic cell transplant (HCT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Histologically confirmed diagnosis of multiple myeloma
* Meeting the Criteria for Symptomatic Multiple Myeloma (CRAB criteria) before the initiation of systemic chemotherapy
* Received high-dose melphalan (≥ 140 mg/m^2) followed by autologous HCT based on the institutional guidelines and within +45 and +180 after autologous HCT at the time of panobinostat maintenance initiation
* Must have achieved at least partial response (PR) prior to autologous HCT and must not have progressive disease (PD) prior to the initiation of maintenance therapy
* Must meet the following laboratory criteria (prior to the initiation of panobinostat maintenance): Absolute neutrophil count (ANC) ≥ 1 x 10^9/L; Hemoglobin ≥ 8 g/dl; Platelets ≥ 50 x 10^9/L (without transfusion support); Creatinine clearance ≥ 40 ml/min or serum creatinine ≤ 2.5 x upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; Serum bilirubin ≤ 1.5 x ULN; Albumin > 3.0 g/dl; Clinically euthyroid. Note: Participants are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Baseline (pre-HCT) multigated acquisition (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥ the limit of normal (LLN) of the institutional normal
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 or Karnofsky performance status ≥ 70%
* Prior histone deacetylase (HDAC), deacetylase (DAC), HSP90 inhibitors or valproic acid for the treatment of cancer is allowed

Exclusion Criteria:

* Potential participants who have purely non-secretory multiple myeloma (i.e., the absence of a measurable protein in serum by electrophoresis and immunofixation and the absence of Bence-Jones protein in the urine defined by use of electrophoresis and immunofixation)
* Prior allogeneic HCT
* Prior solid organ transplant requiring immunosuppressive therapy
* Potential participants who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Impaired cardiac function or clinically significant cardiac diseases
* Diarrhea > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies.
* Have received either immunotherapy within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies
* Have undergone major surgery ≤ 4 weeks prior to starting study drug or have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP must have a negative serum pregnancy test within 24 hours of receiving the first dose of study medication.
* Male patients whose sexual partners are WOCBP not using effective birth control
* A prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiga Nishihori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Relative Dose Intensity (RDI) Per Cohort
Description: Investigators will calculate RDI for each cohort. Relative dose intensity (RDI) represents the ratio of the amount of a drug actually delivered [actual dose intensity (DI)] to the amount planned (planned DI). The purpose of calculating RDI is to evaluate whether the planned DI of a chemotherapy treatment was actually achieved which may suggest the feasibility of planned treatment regimen. There are multitude of reports demonstrating a correlation between RDI and survival in cancer treatment. RDI = (total dose received by the patient = mg)/(planned full dose of drug = mg).
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: percentage of dose
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
Number analyzed (Participants) | 15 | 15
percentage of dose | 97.9 [77.1 to 100] | 89.6 [63.1 to 100]

2. Secondary Outcome: Complete Response Rate
Description: Complete Response (CR) rate to panobinostat maintenance therapy after autologous HCT. CR: Negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
Number analyzed (Participants) | 15 | 15
percentage | 73.33 [44.9 to 92.2] | 66.6 [38.4 to 88.2]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressive Disease (PD) according to Uniform Response Reporting Criteria for Multiple Myeloma by the International Myeloma Working Group (IMWG). Increase of 25% from lowest response value in any of the following:
  * Serum M- component (absolute increase must be ≥ 0.5 g/dL)
  * Urine M-component (absolute increase must be ≥ 200 mg/24 h)
  * Only in patients without measurable serum and urine M protein levels and without measurable disease by free light chain (FLC) levels, bone marrow plasma cell percentage (absolute percentage must be ≥ 10% )
  * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: at 2 years
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
Number analyzed (Participants) | 15 | 15
percentage of participants | 71.8 [41.1 to 88.4] | 53.3 [26.3 to 74.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS: The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Time Frame: at 2 years
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
Number analyzed (Participants) | 15 | 15
percentage of participants | 100 [NA to NA] — first OS event occurred after 24 months | 100 [NA to NA] — first OS event occurred after 24 months

ADVERSE EVENTS:
Time Frame: Adverse events collected from date of consent until off study date, 4 years, 2 months.
Arm/Group | Cohort A: Maintenance Therapy | Cohort B: Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 3/15
Other Adverse Events (participants affected / at risk) | 10/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Maintenance Therapy (N=15) | Cohort B: Maintenance Therapy (N=15)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Maintenance Therapy (N=15) | Cohort B: Maintenance Therapy (N=15)
White blood cell decreased (Investigations) | 6 (14) | 3 (5)
Platelet count decreased (Investigations) | 4 (6) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 5 (5)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 6 (6) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyuria and nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders -Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — bilateral femoral rod placement procedure
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystectomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (7) | 0 (0)
Atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Fibromyalgia (Nervous system disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ottis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT02722941/Prot_SAP_000.pdf